CLINICAL TRIAL: NCT02732444
Title: Erythrocytes Membrane Stability in Chronic Obstructive Pulmonary Disease Patients in Long-Term Home Oxygen Therapy
Brief Title: Erythrocytes Membrane Stability in COPD Patients in Long-Term Home Oxygen Therapy
Status: Completed | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Flaviana Ferreira Gomes, Biologist, Federal University of Uberlandia
Other Study IDs: FUUberlandia 01/2016
Record Dates: First submitted 2016-03-10; First posted 2016-04-08 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Erythrocytes Membranes Stability; Oxidative Stress; Chronic Obstructive Pulmonary Disease (COPD); Advanced Pulmonary Disease (APD); Long-Term Home Oxygen Therapy (LTOT)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD and APD patients in LTOT: • COPD and APD patients in LTOT
- Healthy Control: • Patients without significant cardiorespiratory disease, matched for age and body mass index with the other group.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) patients in Long-Term Home Oxygen Therapy (LTOT) have a reduction in airflow that is not totally reversible. This obstruction may be associated with an abnormal inflammatory response of the lungs as a result of inhalation of toxic particles, particularly to cigarette smoke. Furthermore, COPD patients also present limited symptoms to physical exercise, significant extrapulmonary effects, including weight loss, nutritional abnormalities and skeletal muscle dysfunction. Hyperinflation has been identified as a major cause of dyspnea and is currently believed to be already present in the early stages of the disease, causing limitations in physical capacity. The progressive exertional dyspnea is most associated with impairment to activities of daily living, decreased quality of life and worse prognosis. Traditionally, the severity of COPD is defined by the degree of obstruction, as measured by forced expiratory volume in one second (FEV1) after bronchodilator use (post-BD) and can be classified as mild, moderate, moderately severe and very severe disease. In the group of patients with Advanced Pulmonary Disease (APD), those with partial pressure values of oxygen (PaO2) lower or equal to 55mmHg, or arterial oxygen saturation (SaO2) lower or equal to 88% in ambient air; or those with PaO2 values between 55-60 or SaO2 lower than 90%, with evidence of pulmonary hypertension or polycythemia require LTOT, over 15 hours / day, with evidence of increased survival. The aim of this study is to evaluate the erythrocyte membranes stability in COPD and APD patients in LTOT compared to healthy subjects. It is a cross-sectional, observational study with evaluation of erythrocyte membranes stability among the groups as well as lung function, physical testing, laboratory analysis, oxidative stress and quality of life questionnaires. As red blood cells are the cells responsible for the gas exchange in the lungs and peripheral tissues, and since the patients with COPD and APD have gas exchange impairment compared to the healthy group, it is expected to find a difference in erythrocyte membranes stability and levels of oxidative stress among the groups.

DETAILED DESCRIPTION:
COPD is a major cause of illness and death worldwide, representing a significant economic and social cost. In the household, it causes concern, limited social life and leisure; commits the budget and shortens life. In the professional field, reduces productivity, anticipates the retirement and results in pension payments and benefits. In the area of health system, motivates repeated calls in emergency rooms, outpatient clinics and is a frequent cause of hospitalizations, which causes high costs for government and society. Most cases can be attributed to smoke.

COPD is often developed in middle-aged smokers with long time exposure which have a variety of other diseases related to smoking or aging. COPD itself has also significant extra-pulmonary effects (systemic) that lead to comorbid conditions. Nutritional abnormalities, weight loss and skeletal muscle dysfunction are well-recognized extrapulmonary effects of COPD and patients are at high risk for myocardial infarction, osteoporosis, respiratory infection, bone fractures, depression, sleep disorders, anemia and glaucoma.

Thus, this study aims to investigate the erythrocyte membranes stability in patients with COPD compared to healthy individuals, since the loss or damage of the red blood cells may be related to worsening gas exchange of patients and caused, for example, by increased oxidative stress observed in the disease mechanism of COPD patients, especially those with advanced lung disease.

Cross-sectional, observational study, which will be compared COPD patients with Advanced Lung disease using Long-Term Home Oxygen Therapy to healthy subjects to evaluate the presence of difference in membrane stability in the red blood cells as well as differences in pulmonary function tests, physical tests, laboratory analysis and presence of oxidative stress, as well as their quality of life.

The results obtained after analysis of erythrocyte membranes stability, as well as oxidative stress and functional and laboratory tests will be correlated, both in patients with COPD Long-Term Home Oxygen Therapy as the control group in order to establish relationships between variables and also compare between groups to determine the differences among them.

ELIGIBILITY:
Inclusion Criteria:

1. Control Group

   * Patients without significant cardiorespiratory disease diagnosed, matched for age and body mass index to the group of COPD patients and APD in LTOT;
   * Nonsmoker;
   * Age group over 40 years old;
   * Male gender;
   * Acceptance to participate and agreement to sign the Informed Consent Term
2. COPD Group in LTOT

   * Patients with COPD and APD in LTOT;
   * Patients who do not have associated severe heart disease;
   * Patients with no pulmonary exacerbations in the past four weeks;
   * Male gender;
   * Age group over 40 years old;
   * Acceptance to participate and agreement to sign the Informed Consent Term

Exclusion Criteria:

* Patients with a disability or orthopedic disfunction that unable mobility or performance of physical tests;
* Patients using lipid-lowering drugs such as statins and fibrates;
* Patients or family / guardians who refuse to sign the Informed Consent Term

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Will be selected 100 participants with COPD in Home Oxygen Therapy at HC-UFU, which will be compared with the same amount of healthy individuals, selected in the General Ambulatories of the same hospital and of family health programs of the city of Uberlandia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Erythrocyte Osmotic Fragility Test (FSO) | 1 day
  The stability of erythrocytes is an inverse function of their osmotic fragility and can be measured by erythrocyte osmotic fragility test (FSO). The test of the FSO provides four parameters for the cell stability of measurement: dX, H50, Amax and Amin. Dx parameter expresses variation in salt concentration necessary to take intact erythrocytes (Amin) to a complete lysis state (Amax), with a 100% hemolysis. Increased dX values expresses greater stability of erythrocytes. The H50 parameter is related to the salt concentration required to produce 50% hemolysis. H50 larger values expresses lower stability of erythrocytes.

SECONDARY OUTCOMES:
Blood Sample Collection by venipuncture into test tubes (Vacutainer) containing specific anticoagulants for each dose | 1 day
  The analysis of the following parameters: hematological evaluation (complete blood count), serum levels of folic acid, cobalamin (vitamin B12), homocysteine, lipid profile, lactate dehydrogenase, serum iron, ferritin, transferrin capacity index, uric acid, glucose, albumin, reticulocytes, C-reactive protein (CRP), total bilirubin (TB), direct bilirubin (DB), indirect bilirubin (IB) and glycated hemoglobin (HbA1c).
The blood gases analysis will be performed by Radiometer Copenhagen ABL 330TM device | 1 day
  Will be obtained: potential hydrogen (pH); arterial oxygen tension (PaO2), arterial carbon dioxide tension (PaCO2); and arterial oxyhemoglobin saturation (SaO2). The location and the puncture technique, sample handling and other technical considerations will be made according to the recommendation of specific guidelines of the Brazilian Thoracic Society.
Modified Medical Research Council (MMRC) Dyspnea Scale - Quality of Life Questionnaires | 1 day
  British Medical Research Council developed this scale in order to predict future risk of mortality. The grades vary from 0 to 4, considering 0 better clinical condition and 4 worse health state.
COPD Assessment Test (CAT) - Quality of Life Questionnaires | 1 day
  The CAT consists of eight questions assessing cough, sputum, chest tightness, dyspnea, limitations in home activities, confidence in leaving home, sleep and energy. For each item, the patient chooses only one answer option, whose score ranges from zero to five. At the end of the test, the sum of the scores results in clinical impact of COPD, according to the stratification score of development study and validation of the CAT. The results vary according to the range of the scores, ranked as follows in relation to the clinical impact: 6-10 points, light; 11-20, moderate; 21-30, severe; and 31-40, very serious.
Clinical COPD Questionnaire (CCQ) - Quality of Life Questionnaires | 1 day
  The CCQ is a self-administered questionnaire used routinely for clinical evaluation of COPD patients, but was also accepted as simple and a useful tool to be used in clinical trials evaluating response treatments and interventions. It consists of 10 items that must be answered based on the last seven days of the patient, and the results indicates their clinical condition based on an intensity scale in which zero represents the minimum possible limitation or absence of breathlessness, and six maximum limitation possible. The CCQ has three domains: symptoms, functional status and mental state.
Medical Outcome Study 36-item Short-Form Health Survey (SF-36) - Quality of Life Questionnaires | 1 day
  The SF-36 is a generic tool often used as a measure of health-related quality of life, easy to administer and understand, is composed of 36 items covering eight domains: physical functioning, role limitations due to physical health, pain, general health perception, vitality, social functioning, role limitations due to emotional problems and mental health. It presents a score of 0 (zero) to 100, where zero corresponds to the worst general state of health and 100 corresponds to the best state of health.
St. George's Respiratory Questionnaire (SGRQ) - Quality of Life Questionnaires | 1 day
  The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction. It is self-administered and consists of three domains: symptoms, activity and impact of disease. Each domain has a maximum possible score and the total is expressed as a percentage of that maximum, where values above 10% reflects changes on quality of life. A minimum change in score of 4 units was established as clinically relevant after patient and clinician testing.
Airways questionnaire 20 (Aq-20) - Quality of Life Questionnaires | 1 day
  AQ20 is a specific questionnaire for obstructive respiratory diseases, consisting of only 20 questions, derived from a longer questionnaire: Asthma Quality of Life Questionnaire (AQLQ). On its validation, it was compared to two other more complexes questionnaires (SGRQ and AQLQ) and showed good correlation with these instruments and clinical presentation of the patient. It is self-administered and its great advantage is the short time required to answer it, only 4 minutes, and simplified answers (yes, no or not applicable).

OTHER OUTCOMES:
Spirometry - Pulmonary Function Testing | 1 day
  The spirometric measures pre and post inhalation of 400 µg of salbutamol via metered-dose inhalers will be held in the system Clinical Pulmonary Function-Spirometry. Airflow is measured using a Pitot tube (PreVentPneumotachTM), with flow and volume, and a 3L syringe calibration performed daily, considering the temperature, the humidity and the local barometric pressure. The volunteers completed at least three forced expiratory maneuvers and slow acceptable and at least two reproducible, according to the criteria of the Brazilian Thoracic Society.
Plethysmography - Pulmonary Function Testing | 1 day
  The measurements of static lung volumes will be taken using plethysmography with the Elite Platinum DX system (MGC, Minnesota, USA). Consisting of the following elements: (A) a box with volume of 699 l, that becomes airtight by closing the door; (B) manometer to measure the pressure inside the box; (C) mouthpiece for breathing, consisting of flowmeter by pneumotachography; (D) manometer to measure the pressure in the mouth (equal to alveolar pressure in the absence of airflow and with an open glottis); and (E) of the airflow switch electrically controlled.
Carbon Monoxide Diffusion - Pulmonary Function Testing | 1 day
  DLCO (Carbon Monoxide Diffusion) examine the amount of carbon monoxide (CO) that diffuses from the pulmonary capillaries through alveolar-capillary barrier. The system used for this evaluation will be Platinum Elite DX (MGC, Minnesota, USA), applying the modified Krogh technique (single breath).
Cardiopulmonary Exercise Testing (CPET) In Cycle Ergometry - Physical Tests | 1 day
  The system used is the Cardio 2 (MGC, Minnesota, USA), which consists of a flow module, a gas analyzer and a computer with the software "Breeze Suite 7.2". This controls the ergometer and provides the graphical presentation and examination reports. The gas analyzer determines, breath by breath, the mixed expired fraction of respiratory gases. The analysis of the oxygen (O2) concentration is made using zirconium cell and analysis of the carbon dioxide (CO2) concentration is done in optical analyzer by absorption of infrared light. This module is calibrated before each test, using a reference sample gas (21% of O2 in nitrogen balance) and calibration mixture (12% of O2 and 5% of CO2 in nitrogen balance of the mixture).
Six-Minute Walk Test - Physical Tests | 1 day
  The six-minute walk test (6MWT) is performed in accordance to the American Thoracic Society (ATS) guidelines. The equipment required for the test are: timer, pulse oximeter, heart rate monitor, sphygmomanometer and stethoscope. The tests will be conducted on a 30 meters enclosed corridor, free of obstacles, with chairs positioned at each of its ends, always by the same examiners who will be previously trained. Participants will be instructed to walk as fasten as possible during six minutes, being encouraged with standardized phrases every minute. If necessary, participants can rest, but the timer will remain on and they will be instructed to continue the test as soon as possible until the end of the sixth minute.

CONTACTS AND LOCATIONS:
Overall Officials: Flaviana Gomes, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Hospital of clinics of the federal university of uberlândia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aki H, Yamamoto M. Drug binding to human erythrocytes in the process of ionic drug-induced hemolysis. Flow microcalorimetric approaches. Biochem Pharmacol. 1991 Jan 1;41(1):133-8. doi: 10.1016/0006-2952(91)90021-v. PMID 1986737
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Chasis JA, Mohandas N. Erythrocyte membrane deformability and stability: two distinct membrane properties that are independently regulated by skeletal protein associations. J Cell Biol. 1986 Aug;103(2):343-50. doi: 10.1083/jcb.103.2.343. PMID 3733870
- [Background] Cooper RA. Abnormalities of cell-membrane fluidity in the pathogenesis of disease. N Engl J Med. 1977 Aug 18;297(7):371-7. doi: 10.1056/NEJM197708182970707. No abstract available. PMID 327326
- [Background] Cunha CC, Arvelos LR, Costa JO, Penha-Silva N. Effects of glycerol on the thermal dependence of the stability of human erythrocytes. J Bioenerg Biomembr. 2007 Aug;39(4):341-7. doi: 10.1007/s10863-007-9092-z. Epub 2007 Oct 5. PMID 17917799
- [Background] Finkel T, Holbrook NJ. Oxidants, oxidative stress and the biology of ageing. Nature. 2000 Nov 9;408(6809):239-47. doi: 10.1038/35041687. PMID 11089981
- [Background] McNeil PL, Steinhardt RA. Loss, restoration, and maintenance of plasma membrane integrity. J Cell Biol. 1997 Apr 7;137(1):1-4. doi: 10.1083/jcb.137.1.1. No abstract available. PMID 9105031
- [Background] Montuschi P, Collins JV, Ciabattoni G, Lazzeri N, Corradi M, Kharitonov SA, Barnes PJ. Exhaled 8-isoprostane as an in vivo biomarker of lung oxidative stress in patients with COPD and healthy smokers. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1175-7. doi: 10.1164/ajrccm.162.3.2001063. PMID 10988150
- [Background] Nishimura K, Izumi T, Tsukino M, Oga T. Dyspnea is a better predictor of 5-year survival than airway obstruction in patients with COPD. Chest. 2002 May;121(5):1434-40. doi: 10.1378/chest.121.5.1434. PMID 12006425
- [Background] Park HS, Kim SR, Lee YC. Impact of oxidative stress on lung diseases. Respirology. 2009 Jan;14(1):27-38. doi: 10.1111/j.1440-1843.2008.01447.x. PMID 19144046
- [Background] Penha-Silva N, Firmino CB, de Freitas Reis FG, da Costa Huss JC, de Souza TM, de Freitas MV, Netto RC. Influence of age on the stability of human erythrocyte membranes. Mech Ageing Dev. 2007 Jul-Aug;128(7-8):444-9. doi: 10.1016/j.mad.2007.06.007. Epub 2007 Jun 28. PMID 17681589
- [Background] Singer SJ, Nicolson GL. The fluid mosaic model of the structure of cell membranes. Science. 1972 Feb 18;175(4023):720-31. doi: 10.1126/science.175.4023.720. PMID 4333397
- [Background] Office of the Surgeon General (US); Office on Smoking and Health (US). The Health Consequences of Smoking: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK44695/ PMID 20669512